CLINICAL TRIAL: NCT06966336
Title: IEEM- Work:Rest Cycles in Burn Survivors- Humidity
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Health Resources (Other)
Responsible Party: Principal Investigator, Craig Crandall, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU20250255
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hyperthermia; Burn Injury
Keywords: Burn Survivor; Burn; humid; dry; core temperature; heat; body temperature
MeSH Terms: conditions — Hyperthermia; Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Non-Burned Individuals in Low Humidity Environment: Non-burned individuals will perform up to three work:rest cycles in a heated environment with low humidity, with each work:rest cycle lasting up to 50 minutes.
- Moderate Burned Individuals in Low Humidity Environment: Individuals with moderate sized burn injuries will perform up to three work:rest cycles in a heated environment with low humidity, with each work:rest cycle lasting up to 50 minutes.
- Large Burned Individuals in Low Humidity Environment: Individuals with large sized burn injuries will perform up to three work:rest cycles in a heated environment with low humidity, with each work:rest cycle lasting up to 50 minutes.
- Non-Burned Individuals in High Humidity Environment: Non-burned individuals will perform up to three work:rest cycles in a heated environment with high humidity, with each work:rest cycle lasting up to 50 minutes.
- Moderate Burned Individuals in High Humidity Environment: Individuals with moderate sized burn injuries will perform up to three work:rest cycles in a heated environment with high humidity, with each work:rest cycle lasting up to 50 minutes.
- Large Burned Individuals in HIgh Humidity Environment: Individuals with large sized burn injuries will perform up to three work:rest cycles in a heated environment with high humidity, with each work:rest cycle lasting up to 50 minutes.

SUMMARY:
The purpose of this project is to identify the effects of a severe burn injuries in humans on core temperature responses during work:rest cycles while in a heated environment.

DETAILED DESCRIPTION:
Non-burned control participants and participants who experienced serious burns covering ≥20% of their body surface area will be investigated. Participants will undergo up to three work:rest cycles in the heat (via our environmental chamber) set to no higher than 40 °C. The work:rest cycle will comprise of 30 min of exercise that is followed by up to 20 min of rest, while staying in the heated conditions. Three consecutive work:rest cycles will be performed as illustrated in the protocol document. During one visit, this protocol will be performed in a low humidity state. During the other visit (randomized and crossover), this protocol will be performed in a high humidity state.

ELIGIBILITY:
Inclusion Criteria for Non-burned Individuals:

* Participants must be free of any significant underlying medical problems based upon a detailed medical history and physical exam, and normal resting electrocardiogram. Participants must be between the ages of 18 and 65.

Exclusion Criteria for Non-burned Individuals:

* Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, lung disease, etc.; as well as serious abnormalities detected on routine screening. Current smokers, as well as individuals who regularly smoked within the past 3 years will be excluded. Participants may also be excluded if body mass index is ≥ 31 kg/m2 will likewise be excluded. Participants must not have had a serious burn injury requiring more than 1 night stay in the hospital.

Inclusion Criteria for Individuals with up to 40% of their body surface area burned (moderate burn group):

- Participants must be free of any significant underlying medical problems based upon a detailed medical history and physical exam, and normal resting electrocardiogram. Participants who have sustained a burn injury must have a burn covering 20-40% of their body surface area and 50% of those burns must be full-thickness burns requiring skin grafts. Participants must be between the ages of 18 and 65.

Exclusion Criteria for Individuals with up to 40% of their body surface area burned (moderate burn group):

- Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, lung disease, etc.; as well as serious abnormalities detected on routine screening. Current smokers, as well as individuals who regularly smoked within the past 3 years will be excluded. Participants may also be excluded if body mass index is ≥ 31 kg/m2 will likewise be excluded.

Inclusion Criteria for Individuals with greater than 40% of their body surface area burned (large burn group):

- Participants must be free of any significant underlying medical problems based upon a detailed medical history and physical exam, and normal resting electrocardiogram. Participants who have sustained a burn injury must have a burn covering more than 40% of their body surface area and 50% of those burns must be full-thickness burns requiring skin grafts. Participants must be between the ages of 18 and 65.

Exclusion Criteria for Individuals with greater than 40% of their body surface area burned (large burn group):

- Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, lung disease, etc.; as well as serious abnormalities detected on routine screening. Current smokers, as well as individuals who regularly smoked within the past 3 years will be excluded. Participants may also be excluded if body mass index is ≥ 31 kg/m2 will likewise be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Non-burn control.
  2. Individuals 20 - 40% of their body surface area burned.
  3. Individuals with greater than 40% of their body surface area burned.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in core temperature | From the start of exercise to the end of the last rest period. Approximately at 0 and 170 minutes.
  Change in core body temperature will be measured either from a temperature sensor pill or from a rectal thermometer.

SECONDARY OUTCOMES:
Change in Heart Rate | From the start of exercise to the end of the last rest period. Approximately at 0 and 170 minutes.
  Heart rate will be measured from ECG electrodes attached to the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- IEEM Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No